CLINICAL TRIAL: NCT06566014
Title: Evaluation of XAI-assisted Spina Bifida Diagnosis
Brief Title: The Study Aims to Improve the Accuracy of Detecting Spina Bifida During Early Ultrasound Scans. to Achieve This, an AI Model Has Been Developed to Provide Feedback About the Presence of Spina Bifida. a RCT Has Been Designed to Compare the Effectiveness of AI Feedback with No AI Feedback.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Julie Leth-Petersen, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P-2019-310
Record Dates: First submitted 2024-05-22; First posted 2024-08-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI feedback (Experimental): The participant will receive AI feedback upon completing the task of analyzing 20 images. The AI feedback will include a prediction (Normal/Spina Bifida) along with a confidence score ranging from 0.0 to 1.0, where 0.0 indicates the lowest confidence and 1.0 indicates the highest confidence.
  Interventions: Other: Evaluation of XAI-assisted spina bifida diagnosis
- No AI feedback (Placebo Comparator): The participants will complete the task of analyzing 20 images without any AI feedback.
  Interventions: Other: Evaluation of XAI-assisted spina bifida diagnosis

INTERVENTIONS:
Other: Evaluation of XAI-assisted spina bifida diagnosis — AI feedback

SUMMARY:
The study aims to improve the accuracy of detecting spina bifida during early ultrasound scans. To achieve this, an AI model has been developed to provide feedback about the presence of spina bifida. A RCT has been designed to compare the effectiveness of AI feedback with no AI feedback.

DETAILED DESCRIPTION:
The study aims to improve the accuracy of detecting spina bifida during early ultrasound scans. To achieve this, an AI model has been developed to provide feedback about the presence of spina bifida. A randomized controlled trial (RCT) has been designed to compare the effectiveness of AI feedback with no AI feedback. Forty fetal medicine specialists are randomly assigned to receive either the AI feedback or no feedback, and the two groups are compared to determine if the feedback improved the accuracy of detecting spina bifida.

ELIGIBILITY:
Inclusion Criteria:

* Obstetricians

Exclusion Criteria:

* Fetal medicine specialists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of XAI-assisted spina bifida diagnosis | One month after the survey is distributed.
  The study aims to evaluate whether AI feedback improve the accuracy of diagnosing spina bifida by comparing the number of correct and incorrect responses in a task involving 20 images.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark